CLINICAL TRIAL: NCT01280838
Title: Safer Sex Intervention for Male Clients of Female Sex Workers in Tijuana, Mexico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Thomas L. Patterson, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DA029008
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: HIV; Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Theory-based behavioral intervention (Experimental): Participants in this arm will receive a single-session, theory-based intervention (Hombre Seguro) at baseline that uses principles of behavior change derived from Social Cognitive Theory (SCT), Cognitive Behavioral Therapy (CBT), Theory of Reasoned Action (TRA), and Motivational Interviewing (MI) to increase clients' use of condoms with FSWs. The intervention lasts approximately 45 minutes.
  Interventions: Behavioral: Hombre Seguro
- Didactic attention-control condition (Active Comparator): The didactic control condition is a modified version of the CDC's revised guidelines for HIV counseling, testing, and referral and materials from Mexico's National Center for AIDS Studies (CENSIDA). The one-session, 60-minute counseling intervention focuses on HIV and STI prevention, risk appraisal, and the development of a risk reduction plan.
  Interventions: Behavioral: Didactic attention-control condition

INTERVENTIONS:
Behavioral: Hombre Seguro — A theory-based intervention that uses principles of behavior change derived from Social Cognitive Theory (SCT), Cognitive Behavioral Therapy (CBT), Theory of Reasoned Action (TRA), and MI to increase clients' use of condoms with FSWs.
  Arms: Theory-based behavioral intervention
Behavioral: Didactic attention-control condition — The didactic control condition is a modified version of the CDC's revised guidelines for HIV counseling, testing, and referral and materials from Mexico's National Center for AIDS Studies (CENSIDA). The one-session, 60-minute counseling intervention focuses on HIV and STI prevention, risk appraisal, and the development of a risk reduction plan.
  Arms: Didactic attention-control condition

SUMMARY:
Behavioral interventions designed to reduce risk of HIV and sexually transmitted infections (STIs) have mostly failed to consider clients of female sex workers (FSWs), who may act as a "bridge" to the general population. This study proposes to test a brief, one-hour counseling intervention with male clients in Tijuana, Mexico, to reduce their rates of unprotected sex (i.e., sex without a condom) with FSWs as well as their rates of infection with HIV and STIs. Finding an effective intervention for this population is important given the rising rates of HIV infection in Tijuana (as documented in earlier studies) and the large numbers of people crossing the border in both directions, many of them specifically to purchase sex from FSWs in Tijuana.

DETAILED DESCRIPTION:
Interventions designed to reduce STI/HIV risk have mostly failed to consider clients of FSWs, who may act as a 'bridge' to the general population. Our recent survey of U.S and Mexican clients seeking FSWs in Tijuana revealed a startling HIV prevalence rate of 4.1%. Based on qualitative and quantitative interviews with clients from Tijuana Mexico and the U.S. the investigators developed a theory-based intervention (Hombre Seguro) that uses Motivational Interviewing, active participation, and problem solving to increase clients' use of condoms with FSWs. The investigators now propose an RCT to test the efficacy of this one-hour intervention in Tijuana which will enroll 400 HIV-negative men (200 residents of San Diego County; 200 Tijuana residents) who report having unprotected sex with FSWs in the past 4 months. Our theory-based participatory intervention will be evaluated in comparison with a time and information equivalent didactic control condition. Participants will be recruited in Tijuana where they will undergo a baseline CAPI-administered interview, STI testing (HIV, syphilis, gonorrhea, Chlamydia), and intervention counseling with follow-up interviews at 4, 8, and 12 months post-baseline conducted in either Tijuana or San Diego. Our study aims are to: 1) evaluate the efficacy of Hombres Seguro to increase condom use of clients with FSWs; 2) determine if the intervention is as efficacious among U.S. versus Mexican clients; 3) determine the extent to which theoretically-based components of our intervention (e.g., self-efficacy) represent underlying mechanisms of change in primary outcomes (e.g., lower HIV/STI incidence); and 4) explore subgroup differences in efficacy of the intervention based on background characteristics (e.g., age), contextual factors (e.g., substance use before/during sex), psychosexual factors (e.g., social-sexual effectiveness), and psychosocial factors (e.g., social network influence). Our primary analytic approach will utilize a generalized linear mixed models (GLMM) approach to repeated measures analysis. This bi-national study will contribute significantly to HIV prevention research by addressing the role of male clients in the escalating HIV epidemics in Tijuana and San Diego, and could have application to other settings where HIV prevalence is high among FSWs and their clients.

ELIGIBILITY:
Inclusion Criteria:

* Living in either Tijuana or San Diego County
* Reports having purchased sex for money, drugs, shelter or goods in the last 4 months
* Reports having had unprotected vaginal or anal sex with a FSW in Tijuana at least once during the previous 4 months
* Tests HIV-negative at baseline
* Agrees to receive antibiotic treatment for Chlamydia, gonorrhea, and syphilis if he tests positive (to allow us to differentiate incident from prevalent cases at follow-up)

Exclusion Criteria:

* Consistent use of condoms for vaginal and anal sex with all FSWs during the previous 4 months
* Transgender male (i.e, biologically female)
* Tests HIV-positive at baseline

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of unprotected vaginal or anal sex acts with a female sex worker | 12 months
  Participants will be asked to specify the number of unprotected sex acts they had with female sex workers, spouses, steady partners, and casual partners over the past four months. This question will be asked at baseline and at 4 months, 8 months, and 12 months post-baseline.

SECONDARY OUTCOMES:
HIV status | 12 months
  Participants will be tested for the presence of HIV antibodies at baseline and at 12 months post-baseline.
STI status | 12 months
  Participants will be tested for syphilis, gonorrhea, and chlamydia at baseline and at 12 months post-baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Patterson, Ph.D., Principal Investigator — University of California, San Diego; Carlos Magis Rodriguez, MD, MPH, Study Director — Comisión de Salud Fronteriza Mexico-Estados Unidos
Locations (1):
- Comisión de Salud Fronteriza México-Estados Unidos, Tijuana, Estado de Baja California, Mexico

REFERENCES:
- [Derived] Pitpitan EV, Chavarin CV, Semple SJ, Magis-Rodriguez C, Strathdee SA, Patterson TL. Hombre Seguro (Safe Men): a sexual risk reduction intervention for male clients of female sex workers. BMC Public Health. 2014 May 20;14:475. doi: 10.1186/1471-2458-14-475. PMID 24885949